CLINICAL TRIAL: NCT02662309
Title: A Phase II Study Investigating Preoperative MPDL3280A in Operable Transitional Cell Carcinoma of the Bladder (ABACUS)
Brief Title: Preoperative MPDL3280A in Transitional Cell Carcinoma of the Bladder
Acronym: ABACUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010463QM; 2015-001112-35 (EudraCT Number)
Record Dates: First submitted 2016-01-18; First posted 2016-01-25 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Bladder Cancer
Keywords: Muscle invasive bladder cancer; Transitional cell carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MPDL3280A (Experimental): Patients receive 2x 3-weekly cycles of MPDL3280A (one infusion on the first day of each cycle) prior to cystectomy surgery.
  Interventions: Drug: MPDL3280A

INTERVENTIONS:
Drug: MPDL3280A — Intravenous infusion
  Other Names: Atezolizumab

SUMMARY:
ABACUS is an open-label, international, multi-centre, window of opportunity phase II trial for patients with histologically confirmed (T2-T4a) transitional cell carcinoma of the bladder. The trial aims to test the efficacy of preoperative MPDL3280A and will include extensive biomarker work on samples from these patients. Eligible patients will receive two 3-weekly cycles of MPDL3280A pre-cystectomy. Following cystectomy, patients will be followed up for safety, survival, and disease data.

DETAILED DESCRIPTION:
MPDL3280A (also called atezolizumab) is an immune check point inhibitor which targets programmed death-ligand 1 (PD-L1). Overexpression of PD-L1 prevents the immune system from eradicating cancerous cells as it blocks antigen recognition. MPDL3280A inhibits this interaction, allowing immune-mediated tumour cell killing.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Ability to comply with the protocol
3. Age ≥ 18 years
4. Histopathologically confirmed transitional cell carcinoma (T2-T4a) of the bladder. Patients with mixed histologies are required to have a dominant transitional cell pattern.
5. Residual disease after TURBT (surgical opinion, cystoscopy or radiological presence).
6. Fit and planned for cystectomy (according to local guidelines).
7. N0 or M0 disease CT or MRI (within 4 weeks of registration)
8. Representative formalin-fixed paraffin embedded (FFPE) bladder tumour samples with an associated pathology report that are determined to be available and sufficient for central testing.
9. Patients who refuse neoadjuvant cisplatin based chemotherapy or in whom neoadjuvant cisplatin based therapy is not appropriate.
10. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
11. Negative pregnancy test within 2 weeks of Day 1 Cycle 1 for female patients of childbearing potential.
12. For female patients of childbearing potential to use a highly effecting form(s) of contraception (i.e. one that results in a low failure rate [<1% per year] when used consistently and correctly) and to continue its use for 90 days after the last dose of MPDL3280A.
13. Adequate hematologic and end-organ function within 4 weeks prior to the first study treatment

Exclusion Criteria:

1. Pregnant and lactating female patients.
2. Major surgical procedure within 4 weeks prior to enrolment or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis.
3. Previously intravenous chemotherapy for bladder cancer.
4. Patients with prior allogeneic stem cell or solid organ transplantation.
5. Prior treatment with CD137 agonists, anti-CTLA-4, anti-programmed death-1 (PD-1), or anti-PD-L1 therapeutic antibody or pathway-targeting agents.
6. Patients must not have had oral or IV steroids for 14 days prior to study entry. The use of inhaled corticosteroids, physiologic replacement doses of glucocorticoids (i.e., for adrenal insufficiency), and mineralocorticoids (e.g., fludrocortisone) is allowed.
7. Received therapeutic oral or intravenous (IV) antibiotics within 14 days prior to enrolment (Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible).
8. Administration of a live, attenuated vaccine within 4 weeks prior to enrolment or anticipation that such a live, attenuated vaccine will be required during the study.
9. Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin [IL]-2) within 4 weeks or five half-lives of the drug, whichever is shorter, prior to enrolment.
10. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 4 weeks prior to enrolment.
11. Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome).
12. Malignancies other than UBC within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ treated surgically with curative intent) or localized prostate cancer treated with curative intent and absence of prostate-specific antigen (PSA) relapse or incidental prostate cancer (Gleason score ≤ 3 + 4 and PSA < 10 ng/mL undergoing active surveillance and treatment naive).
13. Severe infections within 4 weeks prior to enrolment in the study including but not limited to hospitalization for complications of infection, bacteraemia, or severe pneumonia.
14. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to enrolment, unstable arrhythmias, or unstable angina.
15. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan (History of radiation pneumonitis in the radiation field (fibrosis) is permitted).
16. Patients with uncontrolled Type 1 diabetes mellitus. Patients with Type 1 diabetes controlled on a stable insulin regimen are eligible.
17. Patients with active hepatitis infection (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
18. Positive test for HIV
19. Patients with active tuberculosis
20. History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug.
21. Uncontrolled hypercalcemia (> 1.5 mmol/L ionized calcium or Ca > 12 mg/dL or corrected serum calcium > the institutional ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab. Patients who are receiving bisphosphonate therapy or denosumab specifically to prevent skeletal events and who do not have a history of clinically significant hypercalcemia are eligible. Patients who are receiving denosumab prior to enrollment must be willing and eligible to receive a bisphosphonate instead while on study.
22. History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
23. Patients with a history of autoimmune-related hypothyroidism, unless on a stable dose of thyroid-replacement hormone.
24. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
25. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the MPDL3280A formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of MPDL3280A pre-cystectomy with respect to pathological complete response rate (pCRR) | 2-3 months (timeframe dependent on delay to surgery)
  Pathological complete response rate defined as no microscopic evidence of residual disease in the bladder based on histological evaluation of the resected bladder specimen collected during cystectomy (post-treatment).

SECONDARY OUTCOMES:
Efficacy of MPDL3280A pre-cystectomy with respect to anti-tumour effects as measured by radiological response (RR) | Approx 34 weeks (timeframe dependent on delay to pre-cystectomy visit)
  CT or MRI scan taken at screening and pre-cystectomy visits. RR is defined as a >30% decrease in tumour diameter from the baseline scan.
Efficacy of MPDL3280A pre-cystectomy with respect to anti-tumour effects based on disease free survival (DFS) | Up to 2 years post-cystectomy
  Disease and survival data is reviewed at post-surgery visits and at 1 and 2 years post-cystectomy.
Efficacy of MPDL3280A pre-cystectomy with respect to anti-tumour effects based on overall survival (OS) | Up to 2 years post-cystectomy
  Disease and survival data is reviewed at post-surgery visits and at 1 and 2 years post-cystectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Powles, MBBS MD MRCP, Principal Investigator — Queen Mary University of London
Locations (20):
- France (4):
  - Centre Hospitalier Universitaire (CHU) de Bordeaux, Bordeaux
  - Hospices Civils de Lyon, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Institut Claudius Régaud, Toulouse
- Netherlands Cancer Institute (NKI), Amsterdam, Netherlands
- Spain (9):
  - Athaia Xarxa Manresa, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Reina Sofía, Córdoba
  - Hospital 12 de Octubre, Madrid
  - CHU de Santiago, Santiago de Compostela
  - Hospital Virgen del Rocío, Seville
- United Kingdom (6):
  - Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton

REFERENCES:
- [Result] Powles, T., et al., A phase II study investigating the safety and efficacy of neoadjuvant atezolizumab in muscle invasive bladder cancer (ABACUS). Journal of Clinical Oncology, 2018. 36(15_suppl): p. 4506-4506.
- [Result] Powles T, Kockx M, Rodriguez-Vida A, Duran I, Crabb SJ, Van Der Heijden MS, Szabados B, Pous AF, Gravis G, Herranz UA, Protheroe A, Ravaud A, Maillet D, Mendez MJ, Suarez C, Linch M, Prendergast A, van Dam PJ, Stanoeva D, Daelemans S, Mariathasan S, Tea JS, Mousa K, Banchereau R, Castellano D. Clinical efficacy and biomarker analysis of neoadjuvant atezolizumab in operable urothelial carcinoma in the ABACUS trial. Nat Med. 2019 Nov;25(11):1706-1714. doi: 10.1038/s41591-019-0628-7. Epub 2019 Nov 4. PMID 31686036
- [Derived] Szabados B, Rodriguez-Vida A, Duran I, Crabb SJ, Van Der Heijden MS, Pous AF, Gravis G, Herranz UA, Protheroe A, Ravaud A, Maillet D, Mendez-Vidal MJ, Suarez C, Linch M, Prendergast A, Tyson C, Mousa K, Castellano D, Powles T. Toxicity and Surgical Complication Rates of Neoadjuvant Atezolizumab in Patients with Muscle-invasive Bladder Cancer Undergoing Radical Cystectomy: Updated Safety Results from the ABACUS Trial. Eur Urol Oncol. 2021 Jun;4(3):456-463. doi: 10.1016/j.euo.2020.11.010. Epub 2021 Feb 18. PMID 33612455